CLINICAL TRIAL: NCT01241305
Title: VCRC Genetic Repository One-Time DNA Protocol
Brief Title: One-Time DNA Study for Vasculitis
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Office of Rare Diseases (ORD) (NIH); Rare Diseases Clinical Research Network (Network)
Responsible Party: Principal Investigator, Peter Merkel, Professor, University of Pennsylvania
Other Study IDs: VCRC5510; U54AR057319-06 (NIH)
Record Dates: First submitted 2010-10-22; First posted 2010-11-16 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Eosinophilic Granulomatosis With Polyangiitis (Churg-Strauss); Giant Cell Arteritis; Granulomatosis With Polyangiitis (Wegener's); Microscopic Polyangiitis; Polyarteritis Nodosa; Takayasu's Arteritis
Keywords: Vasculitis; CSS; EGPA; GCA; GPA; WG; MPA; PAN; TAK
MeSH Terms: conditions — Churg-Strauss Syndrome; Giant Cell Arteritis; Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Polyarteritis Nodosa; Takayasu Arteritis; Vasculitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Two 10 ml tubes of blood will be collected for DNA extraction.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to identify genes that increase the risk of developing vasculitis, a group of severe diseases that feature inflammation of blood vessels. Results of these studies will provide vasculitis researchers with insight into the causes of these diseases and generate new ideas for diagnostic tests and therapies, and will be of great interest to the larger communities of researchers investigating vasculitis and other autoimmune, inflammatory, and vascular diseases.

DETAILED DESCRIPTION:
The systemic vasculitides comprise several inflammatory diseases of blood vessels, usually arteries, which may cause systemic, multi-organ disease that can result in substantial morbidity and increased mortality. Each type of vasculitis is a rare ("orphan") disease. However, taken together, vasculitis affects tens of thousands of Americans and is responsible for substantial morbidity and mortality and almost one billion dollars per year in hospital care alone. While the vasculitides share the trait of vascular inflammation, the unique disease phenotypes, clinical courses, differences in prognoses, and responses to therapy suggest that important differences exist in pathogenesis. The Vasculitis Clinical Research Consortium (VCRC) currently focuses on 6 specific types of vasculitis that were selected to represent a balance between unmet medical and scientific needs, prevalence in North America, feasibility of study, and an interest in studying a spectrum of small, medium, and large vessel vasculitides.

The great majority of published studies on the genetics of vasculitis have used modest-sized cohorts that are only suitable for investigation of a few candidate genes at a time, or to detect large effect sizes, so that replicated findings are highly skewed to the HLA region. Larger and more ambitious genetic studies in vasculitis are expected to generate numerous hypotheses for translational research in gene expression, biochemistry, and molecular pathology.

A one-time collection of clinical data and DNA would substantially increase the sample sizes for genetic association studies in all six vasculitides studied in the VCRC. Many patients are seen at participating VCRC centers but do not enroll in the Longitudinal Studies. These patients often are interested in participating in research studies but cannot return frequently for visits, usually due to distance from the VCRC centers. This approach would be particularly useful for the rarer forms of vasculitis under study (Takayasu's Arteritis (TAK), Polyarteritis Nodosa (PAN), eosinophilic granulomatosis with polyangiitis (Churg-Strauss) (EGPA) and also for Giant Cell Arteritis (GCA), since elderly patients have been particularly likely to decline participation in the Longitudinal Studies due to travel constraints.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnostic criteria for Giant Cell Arteritis Age at disease onset >50 years (required)

1. New onset or new type of localized pain in the head
2. Temporal artery abnormality (i.e. temporal artery tenderness to palpation or decreased pulsation, unrelated to arteriosclerosis of cervical arteries)
3. ESR of >40mm in the first hour by the Westergren method
4. Abnormal artery biopsy (i.e. temporal artery biopsy showing vasculitis characterized by a predominance of mononuclear cell infiltration or granulomatous inflammation, usually with multinucleated giant cells)
5. Large Vessel Vasculitis (LVV) by angiogram or biopsy not explained by something else

Inclusion Criteria:

2. Diagnostic criteria for Takayasu's Arteritis

1. Age at disease onset <50 years
2. Claudication of extremities
3. Decreased brachial artery pulse (one or both arteries)
4. Blood pressure difference of >10mm Hg between the arms
5. Bruit over subclavian arteries or aorta
6. Arteriogram abnormalities compatible with TAK (includes conventional dye angiography or MR angiography or CT angiography)

Inclusion Criteria:

3. Diagnostic criteria for Polyarteritis Nodosa Major criteria (not explained by other causes) felt by investigator to be due to vasculitis

1. Arteriographic abnormality
2. Presence of granulocyte or mixed leukocyte infiltrate in an arterial wall on biopsy
3. Mononeuropathy or polyneuropathy

Minor criteria (not explained by other causes) felt by investigator to be due to vasculitis

1. Weight loss > 4 kg
2. Livedo reticularis, cutaneous ulcerations, or skin nodules
3. Testicular pain or tenderness
4. Myalgias
5. Diastolic blood pressure > 90 mm Hg
6. Elevated BUN or serum creatinine levels
7. Ischemic abdominal pain

Isolated cutaneous Polyarteritis Nodosa 1. Biopsy-proven cutaneous PAN

Inclusion Criteria:

4. Diagnostic criteria for Granulomatosis with Polyangiitis (Wegener's) (GPA) and Microscopic Polyangitis (MPA)

* Diagnosis of GPA or MPA. Widely accepted diagnostic criteria, as opposed to classification criteria or definitions, have not been developed for GPA & MPA.
* For diagnosis of GPA meets at least 2 of the following 5 modified ACR criteria:

  1. Nasal or oral inflammation with oral ulcers or nasal discharge with pus or blood
  2. Abnormal chest radiograph with nodules, fixed infiltrates, or cavities
  3. Urinary sediment with microhematuria or red cell casts
  4. Granulomatous inflammation within the wall of an artery or in the perivascular area on biopsy
  5. Antineutrophil cytoplasmic antibody (ANCA) positive by enzyme immunoassay for either PR3- or MPO-ANCA
* For diagnosis of MPA, meets the Chapel Hill Consensus Conference Definition for MPA:

  1. Necrotizing vasculitis, with few or no immune deposits, that affects small vessels (i.e., capillaries, venules, arterioles)
  2. Necrotizing arteritis involving small- and medium-sized arteries may be present
  3. Necrotizing glomerulonephritis is very common
  4. Pulmonary capillaritis often occurs

     Inclusion Criteria:

     5. Diagnostic criteria for Eosinophilic Granulomatosis with Polyangiitis (Churg-Strauss)
     1. Asthma
     2. Peak peripheral blood eosinophilia of >10% of total WBC
     3. Peripheral neuropathy attributable to vasculitis
     4. Transient pulmonary infiltrates on chest imaging studies
     5. Paranasal sinus abnormalities or nasal polyposis
     6. Eosinophilic inflammation on tissue biopsy

     If patients have 4 of the above 6 criteria but lack clearcut documentation of small vessel vasculitis, they are also eligible for enrollment.

     General Exclusion Criteria:
* Inability to give informed consent and to sign the consent form
* Enrolled in VCRC protocols 5502, 5503, 5504, 5505, 5506, 5522, or 5523
* Unwilling to provide blood for DNA collection

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with giant cell arteritis, Takayasu's arteritis, polyarteritis nodosa, granulomatosis with polyangiitis (Wegener's), microscopic polyangiitis, and eosinophilic granulomatosis with polyangiitis (Churg-Strauss). Enrollment will be sequential and patients will have disease in various stages and of different duration.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-10; Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Evaluation of clinical data and linked DNA specimens. | 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Merkel, MD, MPH, Study Director — University of Pennsylvania
Locations (14):
- United States (11):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Northwestern University, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Hospital for Special Surgery, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
- Canada (2):
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
- Istanbul University, Istanbul, Fatih, Turkey (Türkiye)

REFERENCES:
- [Derived] Doubelt I, Springer JM, Kermani TA, Sreih AG, Burroughs C, Cuthbertson D, Carette S, Khalidi NA, Koening CL, Langford C, McAlear CA, Moreland LW, Monach PA, Shaw DG, Seo P, Specks U, Warrington KJ, Young K, Merkel PA, Pagnoux C. Self-Reported Data and Physician-Reported Data in Patients With Eosinophilic Granulomatosis With Polyangiitis: Comparative Analysis. Interact J Med Res. 2022 May 25;11(1):e27273. doi: 10.2196/27273. PMID 35612893
- See also: Vasculitis Clinical Research Consortium — https://vcrc.rarediseasesnetwork.org/
- See also: Rare Diseases Clinical Research Network — https://www.rarediseasesnetwork.org/